CLINICAL TRIAL: NCT05657691
Title: XanaCIDD: A Double-Blind, Randomized, Placebo Controlled, Parallel-Group Trial to Assess the Safety, Tolerability, and Efficacy of Xanamem® in Adults With Major Depressive Disorder and Impaired Cognition
Brief Title: Xanamem® in Adults With Major Depressive Disorder and Impaired Cognition (XanaCIDD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Actinogen Medical (Industry)
Collaborators: AXIOM Real Time Metrics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACW0008
Record Dates: First submitted 2022-10-17; First posted 2022-12-20 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Major Depressive Disorder; MDD; Cognitive Impairment
Keywords: Xanamem; UE2343; Actinogen; Cortisol; 11β-HSD1; 11-beta-Hydroxysteroid Dehydrogenase Type 1; emestedastat
MeSH Terms: conditions — Depressive Disorder, Major; Cognitive Dysfunction | interventions — UE2343

STUDY DESIGN:
Intervention Model Description: placebo-controlled, parallel-group, double-blind, proof-of-concept trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 10 mg Xanamem™ (Experimental): 10 mg Xanamem™ capsule, to be administered orally once every morning with or without food
  Interventions: Drug: Xanamem™
- Placebo (Placebo Comparator): Placebo capsule, to be administered orally once every morning with or without food
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xanamem™ — Xanamem™ is formulated in green and cream-colored size 3, Coni-Snap-shaped gelatin capsules as an excipient blend at a dose of 10mg. It contains the active pharmaceutical ingredient of UE2343.
  Other Names: UE2343
  Arms: 10 mg Xanamem™
Drug: Placebo — Matching placebo which is identical in appearance to the test product (10 mg Xanamem™ QD) except that it contains no active ingredient.
  Arms: Placebo

SUMMARY:
Xanamem is being developed as a potential treatment for symptomatic, early stages of Alzheimer's Disease (AD) and Major Depressive Disorder (MDD).

This XanaCIDD Phase II study in MDD is to investigate the safety and efficacy of Xanamem™ in treating patients with cognitive and depressive symptoms. Trial participants will be randomized to either receive 10mg of Xanamem™ once daily or a Placebo at a 1:1 ratio in a double-blinded fashion.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female aged 18 to 75, inclusive.
* Positive MDD primary diagnosis confirmed by the Mini-International Neuropsychiatric Interview (MINI).
* Persistent depressive symptoms as determined by a Hamilton Depression Rating Scale (HAM-D) ≥ 17 at Screening.
* Cognitive abilities on a coding test > 0.5 standard deviations below expected.
* Self-reported subjective cognitive dysfunction.
* Currently or previously treated with a stable dose of a first- or second-line antidepressant that is approved for the treatment of depression (but not a tricyclic antidepressant, monoamine oxidase inhibitor, or vortioxetine). If on current treatment, dose must be stable for at least 6 weeks.
* Smokers are eligible if they are able to comfortably abstain from nicotine for 2 hours prior to scheduled cognitive assessments.
* Able to comfortably abstain from caffeine intake for 4 hours prior to scheduled cognitive assessments.
* Must provide written informed consent to participate in the trial and be willing and able to comply with the requirements of the protocol and complete all trial visits.

Key Exclusion Criteria:

* Active suicidal ideation within the previous 3 months
* On a tricyclic antidepressant, monoamine oxidase inhibitor, esketamine, or vortioxetine.
* A history of clinically diagnosed dementia of any type
* Previous clinically significant systemic illness or infection, including test positive COVID-19, within the past 4 weeks prior to Screening
* Has a BMI or body weight that will interfere with participation in the trial
* Type I or Type II diabetes requiring insulin
* Clinically significant ECG abnormalities
* Participation in another clinical trial of a drug or device
* Trial participants who in the opinion of the Investigator exhibit physical, cognitive, or language impairments of such severity as to adversely affect the validity of the data derived from the neuropsychological tests.
* Positive testing for HIV, hepatitis B surface antigen, or hepatitis C antibodies at Screening.
* Participants with a history of drug abuse or addiction in the past 2 years
* Current use of cannabis/marijuana, or tetrahydrocannabinol-containing medications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of Xanamem on attention, including working memory | 6 Weeks (Baseline to Week 6 (end of treatment (EOT)))
  Change from Baseline to EOT in an Attention Composite of a Cognitive Test Battery (CTB) (Detection, Identification, and One Back tests)
Evaluation of the short-term safety and tolerability of Xanamem | 6 Weeks (Baseline to Week 6 (EOT))
  Incidence and severity of treatment-emergent adverse events (TEAEs) Incidence of serious adverse events (SAEs) and SUSARs

SECONDARY OUTCOMES:
Determine the effects of Xanamem on depressive symptoms | 6 Weeks (Baseline to Week 6 (EOT))
  Change from Baseline to EOT on the Montgomery-Åsberg Depression Rating Scale (MADRS).
  The MADRS is a 10-item diagnostic questionnaire used to assess the severity of depressive episodes and is designed to be sensitive to treatment effects. Each item is scored from 0 to 6, and overall scores range from 0 to 60. Higher scores indicate greater severity.

CONTACTS AND LOCATIONS:
Locations (12):
- Australia (7):
  - Paratus Clinical Research Western Sydney, Blacktown, New South Wales
  - Genesis Research Services, Newcastle, New South Wales
  - Paratus Clinical Research Brisbane, Brisbane, Queensland
  - USC Clinical Trials, Sippy Downs, Queensland
  - Ramsay Clinic Albert Road, Melbourne, Victoria
  - Monash Alfred Psychiatry Research Centre, Melbourne, Victoria
  - NeuroCentrix, Noble Park, Victoria
- United Kingdom (5):
  - St Pancras Clinical Research, London
  - Clerkenwell Health, London
  - MAC Clinical Research - Manchester, Manchester
  - Glasgow Memory Clinic, Motherwell
  - MAC Clinical Research - South Yorkshire, Tankersley

REFERENCES:
- See also: Selection and early clinical evaluation of the brain-penetrant 11β-HSD1 inhibitor UE2343 — https://pubmed.ncbi.nlm.nih.gov/28012176/